CLINICAL TRIAL: NCT07007221
Title: Clinical Trials to Evaluate Metformin to Treat Depression in People Living With HIV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDIM-2024-31723
Record Dates: First submitted 2025-03-12; First posted 2025-06-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Depression; Hiv
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome | interventions — Metformin; Fluoxetine

STUDY DESIGN:
Intervention Model Description: This is a 3 part trial, parts 1 and 2 have 2 arms each, part 3 has 4 arms
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1, group 1 (Experimental): HIV patients with depression randomized to metformin dose 1000mg
  Interventions: Drug: Metformin
- Part 1, group 2 (Experimental): HIV patients with depression randomized to metformin dose 1500mg
  Interventions: Drug: Metformin
- Part 2, group1 (Experimental): HIV patients with depression randomized to metformin
  Interventions: Drug: Metformin
- Part 2, group 2 (Placebo Comparator): HIV patients with depression randomized to placebo
  Interventions: Other: Placebo
- Part 3, group 1 (Experimental): HIV patients with depression randomized to Metformin
  Interventions: Drug: Metformin
- Part 3, group 2 (Experimental): HIV patients with depression randomized to fluoxetine
  Interventions: Drug: Fluoxetine
- Part 3, group 3 (Experimental): HIV patients with depression randomized to metformin + fluoxetine
  Interventions: Drug: Metformin+Fluoxetine
- Part 3, group 4 (Experimental): HIV patients with depression randomized to double placebo
  Interventions: Other: double placebo

INTERVENTIONS:
Drug: Metformin — 12 weeks of Metformin 1000mg
  Arms: Part 1, group 1
Drug: Metformin — 12 weeks of Metformin 1500mg
  Arms: Part 1, group 2
Drug: Metformin — 8 weeks of Metformin
  Arms: Part 2, group1
Other: Placebo — 8 weeks placebo drug
  Arms: Part 2, group 2
Drug: Metformin — 12 weeks of Metformin
  Arms: Part 3, group 1
Drug: Fluoxetine — 12 weeks of Fluoxetine
  Arms: Part 3, group 2
Drug: Metformin+Fluoxetine — 12 weeks of Metformin+Fluoxetine
  Arms: Part 3, group 3
Other: double placebo — 12 weeks of double placebo
  Arms: Part 3, group 4

SUMMARY:
Depression in HIV occurs commonly and causes poor HIV outcomes with public health implications.

Depression prevalence in HIV-infected persons is estimated at 26% compared to 5% in the general population. Adherence to antiretroviral medication is a life-saving treatment in HIV, but depression can reduce engagement in care and adherence to medication. Depression is also associated with poorer levels of viral suppression and even mortality. Overall, those with depression and HIV are less likely to return to health and remain more likely to transmit the virus. therefore, treatment of HIV is essential to prevention; lower engagement in and adherence to HIV treatment due to depression puts others at risk. This is a 3 part trial, an initial pilot, a placebo controlled pilot, and a full trial.

Part 1. Dose response, Tolerability/Acceptability of Metformin for Depression in people with HIV: To do Initial assessment of metformin for depression in people with HIV we will perform a randomized, double blind, 2-arm, 12 week randomized controlled trial to assess feasibility and acceptability of metformin for depression. We will test two doses of metformin 1000 mg daily versus 1500 mg daily.

Part 2. Preliminary Efficacy Trial of Metformin for Depression in People with HIV: This will be a two-arm, double-blind trial of metformin versus placebo in people with HIV and depression. We will randomize individuals 1:1 to metformin or placebo. Will then collect blood and rectal swabs for preliminary assessments of the mechanism of action for metformin in people with HIV and depression.

Part 3. Full efficacy factorial trial of metformin for depression and comparison/interaction with fluoxetine in people living with HIV: To assess metformin and fluoxetine as efficacious treatments for depression in people with HIV, we will conduct a 4-arm, 12-week, mechanistic, double-blinded, randomized controlled treatment trial (RCT) with an assessment of inflammation and the gut microbiome. Participants (n=400) will be HIV- positive patients on ART with comorbid depression receiving care at one of two Ugandan clinics. In addition, we will use the NIMH Research Domain Criteria (RDoC) of Acute Threat and loss under Negative Valence using biomarkers and self-reported tools.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* HIV positive
* On HIV antiretroviral therapy for > 6 months
* Undetectable HIV RNA
* Outpatient
* Depression by PHQ-9 >10, confirmed by MADRS score 20+ and MINI interview
* Provision of Informed Consent
* Willingness to comply with all screening and study procedures
* Primary Residence <50 km from clinic

Exclusion Criteria:

* Planning to move out of clinic catchment area in the next 3 months
* Suicidal (PHQ-9 question 9 score >2) or MADRS item 10 with score of 4+
* Pregnant or breastfeeding
* Treatment with a rifamycin
* Current use of any antidepressant, metformin, rifampicin, efavirenz, insulin, or sulfonylurea.
* Active illicit drug use
* Bipolar or psychotic disorder
* Known cirrhosis or heart failure
* Glomerular Filtration Rate (GFR) <45
* Abnormal TSH >3.5 IU/mL
* Previous Enrollment in the trial (Parts 2 and 3)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
MADRS Score | 8 weeks
  A score indicating depression severity, ranging from 0-60 with a higher score indicating more severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lofgren, MD, Principal Investigator — University of Minnesota